CLINICAL TRIAL: NCT04830943
Title: The Effectiveness of Cerebrolycin, a Multi-modal Neurotrophic Factor, for Treatment of Post-covid-19 Persistent Olfactory, Gustatory and Trigeminal Chemosensory Dysfunctions: A Pilot Study
Brief Title: Cerebrolycin for Treatment of Covid-related Anosmia and Ageusia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherifa Ahmed Hamed, Professor of Neurology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-NGF/AUH_SAH/2020
Record Dates: First submitted 2020-12-24; First posted 2021-04-05 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Covid19 Related Anosmia and Aguesia
Keywords: COVID-19; ; anosmia; ; ageusia; ; cerebrolysin
MeSH Terms: conditions — COVID-19; Anosmia; Ageusia | interventions — cerebrolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfactory and gustatory disorders after covid 19 infection (n = 150) (Experimental): Cerebrolysin Dose:5 ml ampoule (1ml contains 215.2 mg cerebrolysin) once daily through intramuscular injection five times per week, for a total of 40 treatments (for at least 8 weeks after presentation), after which the cycle was repeated again according to the each patient response to therapy for a maximum of 24 weeks.
  Interventions: Drug: Cerebrolysin
- control group (n = 100) (No Intervention): no drug intervention, just olfactory training using at least 4 strong odors to smell twice daily for at least 15 minutes (every time), for at least 8 weeks after presentation.

INTERVENTIONS:
Drug: Cerebrolysin — Cerebrolysin will be prescribed in a dose of 5 ml ampoule once daily through intramuscular injection (1ml contains 215.2 mg cerebrolysin) for five times per week, for a total of 40 treatments (for 8 weeks), after which the cycle was individually repeated according to the response of the patient to therapy for a maximum of 24 weeks
  Other Names: Neurotropic factors
  Arms: Olfactory and gustatory disorders after covid 19 infection (n = 150)

SUMMARY:
The loss of smell and taste is a prominent symptom of COVID-19. Studies found that patterns of smell loss due to Covid-19 infection differ from that of other respiratory viruses being much more profound in the Covid-19 patents and did not associate with runny, congested, or blocked-up nose. The researchers suggest that smell and taste testing can be used for fast COVID-19 screening. Studies found that the Covid-19 virus has similarities with severe acute respiratory syndrome coronavirus (SARS-CoV), which has been reported to enter the brain, via smell receptors in the nose. The sudden onset and relatively fast recovery in some patients suggest that COVID-19 anosmia is not caused by damage to the central nervous system but rather by the loss of smell information before it gets to the brain (smell receptors). They also found that it has different behavior from other respiratory viruses as it causes over-reaction of the immune system (or a cytokine storm). Trials to treat post-COVID anosmia using local steroid applications, snifﬁng of strong odors or scents or use of different vitamins (for several weeks to months) did not provide rapid, satisfactory or even significant recovery of olfactory dysfunction. Fortunately, the olfactory neurons can regenerate, however, studies reported variable prognoses, some patients recovered within weeks which others may have persistent deficits for months or even a year. In this study, the researchers hypothesize that cerebrolysin, a drug of neurotrophic and neuroprotective properties, can be used to treat patients with persistent post-COVID anosmia or ageusia or promote functional recovery of smell and taste deficits.

DETAILED DESCRIPTION:
Initial descriptions of the COVID-19 pandemic have focused on its acute severe manifestations. After several months, data have emerged about the mild disease and Post-COVID syndrome. The diminished senses of smell (or hyposmia/anosmia) and taste (or hypogeusia/ageusia) have been commonly reported in the pandemic. Hyposmia/anosmia and hypogeusia/ageusia have also been reported with previous coronaviruses. In late March, the professional society of Ear, Nose, and Throat (ENT) in the United Kingdom (UK) published an advisory on evidence from South Korea, China, and Italy that signiﬁcant number of COVID-19 positive patients also lost smell and/or taste. Based also on several other reports which reported that 66-88% of patients have lost smell and/or taste due to COVID-19 infection, the American Academy of Otolaryngology-Head and Neck Surgery and World Health Organization (WHO) have added anosmia and ageusia to the list of symptoms of COVID-19. The prognosis of such deficits seems variable. Some reported recovery within few weeks; while many reported persistence of deficits for several months or even more than a year after the onset of the condition. Furthermore, some patients developed respiratory symptoms later after anosmia while others remained asymptomatic. The exact mechanisms for these deficits are still under research. In animal models, the investigators found that coronaviruses could impair the olfactory neuroepithelium through the expression of angiotensin-converting enzyme type 2 (ACE2) in the sustentacular cells or damage the receptors. Treatment trials of post-COVID anosmia included the application of nasal corticosteroids, regular snifﬁng of different odors and strong scents, and treatment with antioxidants and vitamins or interventions as olfactory training. However, none was therapeutically effective. Previous preclinical and clinical studies have shown that treatment with neurotrophic polypeptides can promote neurological recovery for many neurodegenerative and acquired nervous system diseases due to different causes. As the olfactory neurons are capable of regeneration, the researchers propose that treating patients with prolonged post-COVID anosmia or ageusia using cerebrolysin, a drug of neurotrophic and neuroprotective properties may promote recovery of olfactory and gustatory dysfunctions. Cerebrolysin is a mixture of peptides purified from brains, including (and not limited to) brain-derived neurotrophic factor (BDNF), glial cell line-derived neurotrophic factor (GDNF), nerve growth factor (NGF), and ciliary neurotrophic factor (CNTF).

ELIGIBILITY:
Inclusion Criteria:

* A random sample of at least 250 adults with sudden hyposmia/anosmia and/or hypoageusia/ageusia during COVID-19 pandemics and experienced persistent olfactory and/or gustatory manifestations after recovery from other acute viral manifestations.
* compliance for drug intervention (group 1) or olfactory training (group 2) for at least 8 weeks.

Exclusion Criteria:

* Prior neurologic, medical or psychiatric disease.
* Other known infection at onset
* Nasal congestion
* Nasal polyps
* Surgery or head trauma or radiation for head and neck cancers as may result in injury to the nerves that control smell
* Exposure to toxic chemicals (such as pesticides and solvents)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The smell and taste questionnaire component of the National Health and Nutrition Examination Survey (NHNES). And the modified Arabic translated and validated sniffin' sticks odor identification test was used for objective olfactory evaluations. | The subject smell and taste sensations at baseline (presentation)
  The NHNES questions have been selected to characterize the variation, timing and associated-symptoms of both olfactory and gustatory systems.
objective testings: sniffen's odor, taste and flavor identification testing | at presentation (baseline)
  For quantitative assessment of smell, we used 16 odors familiar to Egyptians For quantitative assessment of taste loss, we used sugar (sweet), salt (salty), lemon (sour), old rumi cheese chips (umami) and coffee (bitter), the five basic tastants.
  For quantitative assessment of flavor, we used 16 recipes familiar for Egyptians.

SECONDARY OUTCOMES:
The Globas Rating for smell (GRS) | 8 weeks, 12 weeks, 16 weeks, 18 weeks and 24 weeks
  GRS is a single-item, global rating that asks the patient to rate his current sense of smell as follow: excellent, very good, good, fair, poor or absent
The Globas Rating for taste (GRT) | 8 weeks, 12 weeks, 18 weeks and 24 weeks
  GRT is a single-item, global rating that asks the patient to rate his current sense of taste as follow: excellent, very good, good, fair, poor or absent
objective testings: sniffen's odor, taste and flavor identification testing | at 8, 12, 16, 18 and 24 weeks after intial evaluation at baseline
  For quantitative assessment of smell, we used 16 odors familiar to Egyptians For quantitative assessment of taste loss, we used sugar (sweet), salt (salty), lemon (sour), old rumi cheese chips (umami) and coffee (bitter), the five basic tastants.
  For quantitative assessment of flavor, we used 16 recipes familiar for Egyptians.

CONTACTS AND LOCATIONS:
Overall Officials: Sherifa A Hamed, M.D., Principal Investigator — Assiut University, Faculty of Medicine
Locations (1):
- Assiut University Hospitals, Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chachkhiani D, Soliman MY, Barua D, Isakadze M, Villemarette-Pittman NR, Devier DJ, Lovera JF. Neurological complications in a predominantly African American sample of COVID-19 predict worse outcomes during hospitalization. Clin Neurol Neurosurg. 2020 Oct;197:106173. doi: 10.1016/j.clineuro.2020.106173. Epub 2020 Aug 25. PMID 32877769
- [Background] Shrestha GS, Khanal S, Sharma S, Nepal G. COVID-19: Current Understanding of Pathophysiology. J Nepal Health Res Counc. 2020 Nov 13;18(3):351-359. doi: 10.33314/jnhrc.v18i3.3028. PMID 33210623
- [Background] Veinbergs I, Mante M, Mallory M, Masliah E. Neurotrophic effects of Cerebrolysin in animal models of excitotoxicity. J Neural Transm Suppl. 2000;59:273-80. doi: 10.1007/978-3-7091-6781-6_29. PMID 10961439
- [Result] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535
- [Derived] Hamed SA, Ahmed MAA. The effectiveness of cerebrolysin, a multi-modal neurotrophic factor, for treatment of post-covid-19 persistent olfactory, gustatory and trigeminal chemosensory dysfunctions: a randomized clinical trial. Expert Rev Clin Pharmacol. 2023 Jul-Dec;16(12):1261-1276. doi: 10.1080/17512433.2023.2282715. Epub 2023 Dec 9. PMID 37950370